CLINICAL TRIAL: NCT05367609
Title: Personalized Perioperative Analgesia Platform (PPAP) for Pediatric Spine Fusion Surgery (sIRB)
Acronym: PPAP Spine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Senthil Sadhasivam (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Senthil Sadhasivam, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21090075; TR003719 (Other Grant/Funding Number: National Institutes of Health)
Record Dates: First submitted 2022-04-19; First posted 2022-05-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: PPAP; Spine Fusion
Keywords: PPAP; Pediatric; Spine Fusion Surgery

STUDY DESIGN:
Intervention Model Description: PK sampling and genetic testing will determine the type of analgesia medication treatment the patient receives
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Children undergoing Spine Fusion Surgery (Other): This arm will include approximately 300 children undergoing spine fusion surgery
  1. Pharmacokinetic (PK): collection of 10-13 serial blood samples to determine serum levels of methadone/oxycodone and its metabolites
  2. Pharmacogenetic (PG): Preoperative CYP2D6 genotyping (for preferential recruitment of CYP2D6 PMs and UMs). This will be collected in the pre-operative clinic via blood if there are clinical labs needed for standard of care. If no blood is needed in the pre-op clinic, the investigators will collect this via saliva.
  Postoperative Analgesia Dose and PK Sampling Schedule:
  Clinical care providers are blinded to CYP2D6/CYP2B6 when prescribing oxycodone/methadone; and genetic analysis of proposed targeted genes. Results of these samples will be used to determine personalized analgesia plan.
  Interventions: Diagnostic Test: Preoperative Genotyping

INTERVENTIONS:
Diagnostic Test: Preoperative Genotyping — Genotype based risk prediction and personalized pain management

SUMMARY:
The purpose of this collaborative CTSA application is to develop an innovative perioperative precision analgesia platform (PPAP) to improve analgesia and reduce serious immediate and long-term adverse outcomes of perioperative opioids in children undergoing painful surgery.

DETAILED DESCRIPTION:
Aim 1. Develop and implement a perioperative precision analgesia platform (PPAP) by linking genomics to opioid metabolism, CPIC guidelines, precision dosing, clinical safety, and personalizing analgesia

Aim 2. Implement and evaluate PPAP in children undergoing major inpatient surgery, posterior spinal fusion (PSF)

1. Determine genetic factors predisposing children to immediate and long-term postoperative methadone and oxycodone related adverse effects including RD, PONV, opioid dependence, and CPSP The investigators postulate that specific CYP2B6, ABCB1, OPRM1, FAAH, and CYP2D6 variants identify children at risk for poor pain relief, RD, PONV, opioid dependence, and CPSP in the postoperative period.
2. Determine genetic variants-based perioperative dosing and outpatient prescribing of opioids

The investigators hypothesize that CYP2B6 and CYP2D6 variants will explain pharmacokinetic variations of methadone and oxycodone, determine the right doses, and implement precision opioid use for optimal clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

* Children ages 10 to 21
* ASA physical status 1 to 3
* Undergoing Posterior-Lateral Spinal Fusion
* Receives in-patient opioids
* Prescribed opioids at discharge

Exclusion Criteria:

* Serious illness
* Preoperative severe pain
* Preoperative opioid use or misuse

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Look at genetic factors predisposing children to immediate postoperative opioid-adverse effects Respiratory Depression (RD) and Postoperative Nausea and Vomiting (PONV) | Immediately post-surgery
  The investigators will look at specific CYP2D6, ABCB1, FAAH, OPRM1, and COMT variants to find correlations with children who experience RD and PONV in the immediate post-surgical period (4 days) in the hospital
Look at genetic factors predisposing children to postoperative opioid-adverse effects Respiratory Depression (RD) and Postoperative Nausea and Vomiting (PONV) at genetic factors predisposing children to inadequate surgical pain relief with oxycodone | At home up to 1 year post-surgery
  The investigators will look at specific CYP2D6, ABCB1, FAAH, OPRM1, and COMT variants to find correlations with children who experience RD and PONV in the post-surgical period at home up to 1-year
Look at genetic factors predisposing children to inadequate surgical pain relief with oxycodone | Immediately post-surgery
  The investigators will look at specific CYP2D6, ABCB1, FAAH, OPRM1, and COMT variants to find correlations with children who experience poor pain relief in the immediate post-surgical period (4 days) in the hospital. Poor pain relief will be determined using the Numerical Rating Scale (NRS) which runs on a 0-10 scale; 0 being no pain at all, 10 being the worst pain imaginable.
Look at genetic factors predisposing children to inadequate surgical pain relief with oxycodone | At home up to 1 year post-surgery
  The investigators will look at specific CYP2D6, ABCB1, FAAH, OPRM1, and COMT variants to find correlations with children who experience poor pain relief in the post-surgical period at home up to 1-year. Poor pain relief will be determined using the Numerical Rating Scale (NRS) which runs on a 0-10 scale; 0 being no pain at all, 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Look at the impact of CYP2D6 variants on oxycodone's clinical dosing in children to see if specific variants correlate with a need for lower or higher doses of analgesic | Pre-operative to post-operative day 2
  The investigators will look at CYP2D6 variants to find correlations in oxycodone's PK sampling and the need for dose adjustments that lead to desired clinical outcomes in children undergoing major inpatient surgeries. Oxycodone will be measured by the IU CTSI's Clinical Pharmacology Analytical Core (CPAC) laboratory using a validated LC/MS/MS as-say,201 and plasma alpha-1 acid glycoprotein (AAG) will be measured using a HPLC/UV assay. Study team will track the subjects choices from their signed consent form regarding PK collections.

OTHER OUTCOMES:
Look at OPRM1 epigenetics and OPRM1, FAAH, GCH1, DRD2 variants to find correlations with chronic persistent surgical pain (CPSP) up to 1-year post-surgery | Post-operative up to 1-year
  Children will be asked to complete psychological questionnaires post-surgery to assess psycho-psychological factors that may correlate with CPSP. CPSP is defined as pain that develops after a surgical procedure and lasts at least 3 months and significantly affects health-related quality of life.
Look at OPRM1 epigenetics and OPRM1, FAAH, GCH1, DRD2 variants to find correlations with opioid dependence (OD) up to 1-year post-surgery | Post-operative up to 1-year
  Children will be asked to complete psychological questionnaires post-surgery to assess psycho-psychological factors that may correlate with opioid dependence (OD). OD will be determined using the validated Sophia Observation Withdrawal Symptoms Scale and the Clinical Opiate Withdrawal Scale (COWS). The Sophia Observation Withdrawal Symptoms Scale is based on a 15-point scale. The COWS is based on a scale with a minimum score of 5 and maximum score of 48; 5-12 = mild, 13-24 = moderate, 25-36 = moderately severe, more than 36 = severe withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Senthilkumar Sadhasivam, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - University of California, San Francisco, California
  - Riley Children's Hospital, Indianapolis, Indiana
  - UPMC Children's Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No current IPD sharing plan anticipated